CLINICAL TRIAL: NCT03535883
Title: The Safety of Thoracentesis, Tunneled Pleural Catheter (Pleurx), and Chest Tubes in Patients Taking Novel Oral Anti-Coagulants (NOAC).
Brief Title: The Safety of Thoracentesis, Tunneled Pleural Catheter, and Chest Tubes in Patients Taking Novel Oral Anti-Coagulants
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 2000021542; No NIH funding (Other: 10.11.23)
Record Dates: First submitted 2018-05-08; First posted 2018-05-24 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Pleural Effusion; Thoracic Effusion
MeSH Terms: conditions — Pleural Effusion | interventions — N(4)-oleylcytosine arabinoside

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients taking NOAC's: Patients with unilateral or bilateral pleural effusions who undergo thoracentesis, chest tube, or pleurx placement and are taking Novel Oral Anti-Coagulants (NOAC).
  Interventions: Drug: Novel Oral Anti-Coagulants
- patients not taking NOAC's: Patients with unilateral or bilateral pleural effusions who undergo thoracentesis, chest tube, or pleurx placement who are not taking Novel Oral Anti-Coagulants (NOAC).

INTERVENTIONS:
Drug: Novel Oral Anti-Coagulants — Novel Oral Anti-Coagulant (NOAC) medications (i.e. Eliquis, Plavix, Xarelto etc.)
  Other Names: NOAC
  Groups: patients taking NOAC's

SUMMARY:
To assess risks of bleeding in those individuals receiving Novel Oral Anti-Coagulant (NOAC) medications, admitted to the hospital and require thoracentesis, chest tube or tunneled pleural catheter placement.

DETAILED DESCRIPTION:
The research component of this study simply observes and documents the outcomes of these procedures. Patients will undergo an analysis of their pre-procedural hematocrit and this will be compared to their post-procedural (next day) hematocrit.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 y/o
2. Unilateral or bilateral pleural effusion
3. Ability to provide consent or consent given for the procedure and research study

Exclusion Criteria:

Adults who refuse to provide consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with unilateral or bilateral pleural effusions who undergo thoracentesis, chest tube, or pleurx placement.
Sampling Method: Non-Probability Sample
Enrollment: 590 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Risk of bleeding | 2 years
  Reduced risk of bleeding in individuals receiving Novel Oral Anti-Coagulants as well as those that are in the control group will be assessed by having the patients undergo an analysis of their pre-procedural hematocrit which will be compared to their post procedural (next day) hematocrit

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Bramley, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States